CLINICAL TRIAL: NCT01902472
Title: A Prospective, Observational Study of Individuals Who Seroconvert While Taking Truvada® for Pre-Exposure Prophylaxis (PrEP)
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-US-276-0103; EUPAS24374 (Registry Identifier: ENCePP)
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: HIV
Keywords: HIV-1; Truvada; FTC/TDF; Pre-exposure prophylaxis; PrEP; Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- FTC/TDF for PrEP: HIV-1 negative adults (any sex/gender, including transgender) who seroconvert while taking FTC/TDF for PrEP

SUMMARY:
This study will evaluate HIV-1 RNA and the presence or absence of resistance at baseline and following seroconversion, assess the frequency of HIV-1 screening and screening method(s) used for evaluation of seroconverters, and collect information regarding whether the seroconverter experienced signs and symptoms of acute HIV-1 infection prior to or at the time of seroconversion.

ELIGIBILITY:
Inclusion Criteria:

* Participant in a FTC/TDF PrEP demonstration project or FTC/TDF for PrEP clinical study
* HIV-1 negative adults (any sex/gender, including transgender) ≥ 18 years of age at time of enrollment in the demonstration project or clinical study.
* Evidence of seroconversion while receiving FTC/TDF for PrEP

Exclusion Criteria:

* This is an observational nested study and will monitor all reported seroconversions without intervention/exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred fifty (150) HIV-1 negative adults (any sex/gender, including transgender) and ≥ 18 years of age who seroconvert while taking FTC/TDF for PrEP.
Sampling Method: Non-Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2013-09-02 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate among all subjects exposed to emtricitabine (FTC)/ tenofovir disoproxil fumarate (TDF) (Truvada®) for a PrEP indication | Baseline to Year 3
Proportion of seroconverters with resistance mutations | Baseline to Year 3
Proportion of seroconverters with signs/symptoms at or before seroconversion | Baseline to Year 3

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Inc., Foster City, California, United States

IPD SHARING:
Plan to Share IPD: No